CLINICAL TRIAL: NCT07369336
Title: Clinical Outcomes of Inhaled Amikacin in Ventilator Associated Pneumonia:A Group Randomized Controlled, Add on Trial
Brief Title: Clinical Outcomes of Inhaled Amikacin in Ventilator Associated Pneumonia
Acronym: RCT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Postgraduate Medical Institute, Lahore (Other)
Responsible Party: Principal Investigator, Anum Anwar, Assistant Professor Anaesthesia/ICU, Postgraduate Medical Institute, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LGH/PGMI/AMC
Record Dates: First submitted 2025-12-08; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: Ventilator associated pneumonia; Inhaled amikacin; Mechanical ventilation; Adjunctive therapy; Clinical improvement
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Amikacin; Inhalation

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two independent parallel groups.One group received standard empirical therapy ie. intravenous antibiotics, while the other group received inhaled amikacin in addition to same intravenous antibiotic regimen. Both groups were treated concurrently without crossover, allowing direct comparison of clinical outcomes between the two treatment strategies.
Masking Description: No masking was applied. Due to nature of treatmeht, both the treating clinicians and participants, representatives were aware of the assigned treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhaled Amikacin + Standard-of-Care Antibiotics (Experimental): Participants will receive inhaled amikacin administered via nebulization in addition to standard intravenous antibiotic therapy for ventilator-associated pneumonia. Therapy continues for the prescribed antibiotic course and according to unit protocol.
  Interventions: Drug: Amikacin (Inhalation); Drug: Standard-of-Care Intravenous Antibiotics
- Participants will receive ONLY standard of care antibiotics (Active Comparator): Participants will receive only standard intravenous antibiotic therapy for ventilator-associated pneumonia. Therapy continues for the prescribed antibiotic course and according to unit protocol.
  Interventions: Drug: Standard-of-Care Intravenous Antibiotics

INTERVENTIONS:
Drug: Amikacin (Inhalation) — Amikacin administered as an aerosolized solution via a vibrating mesh nebulizer once daily for the duration of systemic antibiotic therapy, according to ICU protocol for ventilator-associated pneumonia.
  Arms: Inhaled Amikacin + Standard-of-Care Antibiotics
Drug: Standard-of-Care Intravenous Antibiotics — Intravenous antibiotics selected based on local antimicrobial guidelines and pathogen sensitivity for ventilator-associated pneumonia, administered for the full

SUMMARY:
Article: Clinical Outcomes of Inhaled Amikacin in Ventilator-Associated Pneumonia: A group randomized controlled,add-on trial English:Patients in intensive care units often need ventilators to breathe. Sadly, these machines sometimes cause serious lung infections, known as ventilator-associated pneumonia (VAP). This study tested whether giving the antibiotic amikacin by inhalation (so itgoes straight into the lungs) could improve recovery when added to regular treatment. Researchers looked at how quickly infections cleared, how long patients needed the ventilator, and whether hospital stays were shortened. They also monitored for side effects.

DETAILED DESCRIPTION:
Ventilator-associated pneumonia continues to pose a significant therapeutic challenge due to rising antimicrobial resistance and suboptimal lung penetration of systemic antibiotics. Inhaled amikacin offers the advantage of delivering high local drug concentrations in the respiratory tract with minimal systemic toxicity.

This group randomized controlled add-on trial was conducted in the Surgical Intensive Care Units of Lahore General Hospital, Pakistan, from January to December 2024. A total of 180 adult patients diagnosed with VAP were allocated to one of two treatment arms:

Group N (Control): Empirical intravenous antibiotics (Meropenem ± Moxifloxacin)

Group A (Intervention): Inhaled amikacin (20 mg/kg/day in two divided doses) in addition to empirical intravenous antibiotics

Randomization was computer-generated and stratified by age, gender, and baseline SOFA score.

Clinical outcomes assessed included fever resolution, leukocyte normalization, reduced oxygen requirement, radiographic improvement, ventilator weaning, duration of mechanical ventilation, and length of ICU stay. Composite clinical improvement was defined as improvement in at least three out of five predefined domains.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

Participants must meet all of the following:

1. Age 18-80 years
2. Currently receiving invasive mechanical ventilation
3. Clinical diagnosis of ventilator-associated pneumonia (VAP) based on:

   New or progressive infiltrate on chest imaging and at least two of the following:

   Fever > 38°C or hypothermia < 36°C

   Leukocytosis >12,000 or leukopenia <4,000 cells/µL

   Increased purulent respiratory secretions

   Worsening oxygenation indices
4. Initiation of systemic IV antibiotics for VAP
5. Availability of baseline respiratory sample for culture
6. Informed consent obtained from patient's legal guardian/attendantExclusion Criteria

Any of the following will lead to exclusion:

1. Known hypersensitivity to aminoglycosides (e.g., amikacin)
2. Chronic kidney disease Stage 4-5 or baseline serum creatinine >2 mg/dL
3. Pre-existing hearing loss or vestibular dysfunction
4. Severe bronchospasm or airway instability preventing safe nebulization
5. VAP due to confirmed pan-resistant microorganisms requiring alternative therapy

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Duration of invasive mechanical ventilation | From randomization until successful discontinuation of mechanical ventilation, assessed up to 28 days
  The total number of consecutive days a participant remains on invasive mechanical ventilation following enrollment. Extubation is considered successful if the participant remains off the ventilator for at least 48 hours without the need for reintubation.

SECONDARY OUTCOMES:
Clinical Improvement on Day 7 | Day 7 after initiation of study treatment
  The proportion of participants achieving a predefined composite improvement in clinical status, including:
  Reduction in sputum volume and purulence
  Reduction in requirement for oxygen support
  Improvement in PaO₂/FiO₂ ratio
  Radiological improvement on chest imaging
  Resolution of fever (temperature <38°C for >24 hours)
  Measured using standardized clinical criteria for ventilator-associated pneumonia.

CONTACTS AND LOCATIONS:
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in this article may be shared upon reasonable request from qualified researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months after publication of study results, with no planned end date.
Access Criteria: Requests must include a methodologically sound proposal and will require approval by the Institutional Review Committee and execution of a data sharing agreement.
URL: https://sites.google.com/view/inhaled-amikacin-vap-data

REFERENCES:
- See also: https://sites.google.com/view/inhaled-amikacin-vap-data — https://www.mattioli1885journals.com/index.php/actabiomedica/article/view/13910

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-01-03): https://cdn.clinicaltrials.gov/large-docs/36/NCT07369336/Prot_SAP_ICF_000.pdf